CLINICAL TRIAL: NCT01379976
Title: Randomized, Double-blind, Placebo-controlled Phase 3 Trial to Assess the Efficacy and Safety of Acetyl-L-carnitine in Combination With a Cisplatin-containing Chemotherapy as First Line Treatment of Advanced or Metastatic Non Small Cell Lung Cancer
Brief Title: Acetyl-L-carnitine in Combination With a Cisplatin-containing Chemotherapy as First Line Treatment of Advanced or Metastatic Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment was prematurely stopped due to difficulty of recruitment encountered by the experimental centers
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-022021-15
Record Dates: First submitted 2011-06-16; First posted 2011-06-23 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung; cancer; non small cell lung cancer; Advanced or metastatic non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHT cisplatin containing + placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CHT cisplatin containing + acetyl-L-carnitina (Experimental)
  Interventions: Drug: Acetylcarnitine

INTERVENTIONS:
Drug: Acetylcarnitine — ALC or placebo will be administered concurrently with CHT at 1000 mg sachet three times every day (before meals).
  Treatment should be administered for a maximum of 6 cycles for both arms unless progression or unacceptable toxicity, or treatment refusal.
  Other Names: ST 200
  Arms: CHT cisplatin containing + acetyl-L-carnitina
Drug: Placebo — ALC or placebo will be administered concurrently with CHT at 1000 mg sachet three times every day (before meals).
  Treatment should be administered for a maximum of 6 cycles for both arms unless progression or unacceptable toxicity, or treatment refusal.
  Arms: CHT cisplatin containing + placebo

SUMMARY:
Study objectives Primary: To compare toxicity free survival of patients treated with ALC (acetylcarnitine) plus cisplatin-containing chemotherapy (CHT) versus those treated with placebo plus cisplatin-containing chemotherapy.

Secondary: To compare progression free survival, overall survival, the compliance to treatment, the number of episodes of grade 3-4 National Cancer Institute Common Terminology Criteria for Adverse Events, version 3.0, neurotoxicity, as well as the proportion of patients experiencing grade 2-3-4 National Cancer Institute Common Terminology Criteria for Adverse Events, neuropathic pain intensity, the clinical signs and/or symptoms (such as burning, numbness, itching, etc.) of the sensorial neuropathy between the two treatment arms. Study design Multicentre, randomised, double-blind, placebo-controlled, phase III, superiority study in patients with advanced or metastatic NSCLC (non small cell lung cancer).

Patients to be screened for study inclusion are those for which the decision to start a cisplatin-containing treatment has been already taken in the context of the clinical practice. The type of cisplatin-based treatment is not fixed, but each single investigator is free to choose for each single patient among those already approved for first line treatment of advanced or metastatic NSCLC.

Patients meeting the eligibility criteria will be randomized with a 1 : 1 ratio to receive ALC + cisplatin-containing CHT or Placebo + cisplatin-containing CHT until patient refusal, disease progression, unacceptable toxicity or death. The study will be conducted in Italy in approximately 20 investigational centers in order to recruit 650-675 subjects over a 30-month period.

Both efficacy and safety data will be collected. Follow-up will be according to the clinical practice. Data capture will continue, for each patient, until death or study closure.

DETAILED DESCRIPTION:
Inclusion criteria:

* Male or female >= 18
* No previous CHT or targeted therapies. Previous adjuvant or neo-adjuvant treatment is permitted if completed ≥ 6 months before study inclusion.
* ECOG performance status 0-1
* Adequate organ functions defined as follows:
* Neutrophils >= 1.5 x 109/L, platelets >= 100 x 109/L, and hemoglobin >= 9 g/dL
* Bilirubin level either normal or < 1.5 x ULN
* ASAT and ALAT <= 2.5 x ULN (<= 5 x ULN if liver metastasis are present)
* Serum creatinine <1.5 x ULN
* Written informed consent given before the randomization, according to International Conference on Harmonization/Good Clinical Practice (ICH/GCP)

Exclusion criteria:

* Symptomatic brain metastases
* Any investigational agent(s) within 4 weeks prior to study entry
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease
* Patients with known allergy to any other components of the study drugs
* History or presence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or patient at high risk from treatment complication
* Known drug abuse/ alcohol abuse
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent
* Clinically relevant peripheral neuropathy
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix (Patients with a previous malignancy but without evidence of disease for 5 years will be allowed to enter the trial)
* Pregnancy or breast feeding. Women of childbearing potential and their parents must be willing to practice acceptable methods of birth control to prevent pregnancy
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18
* No previous CHT or targeted therapies. Previous adjuvant or neo-adjuvant treatment is permitted if completed ≥ 6 months before study inclusion.
* ECOG performance status 0-1
* Adequate organ functions defined as follows:
* Neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, and hemoglobin ≥ 9 g/dL
* Bilirubin level either normal or < 1.5 x ULN
* ASAT and ALAT < 2.5 x ULN (< 5 x ULN if liver metastasis are present)
* Serum creatinine <1.5 x ULN
* Written informed consent given before the randomization, according to International Conference on Harmonization/Good Clinical Practice (ICH/GCP)

Exclusion Criteria:

* Symptomatic brain metastases
* Any investigational agent(s) within 4 weeks prior to study entry
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease
* Patients with known allergy to any other components of the study drugs
* History or presence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or patient at high risk from treatment complication
* Known drug abuse/ alcohol abuse
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent
* Clinically relevant peripheral neuropathy
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix (Patients with a previous malignancy but without evidence of disease for < 5 years will be allowed to enter the trial)
* Pregnancy or breast feeding. Women of childbearing potential and their parents must be willing to practice acceptable methods of birth control to prevent pregnancy
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Toxicity Free Survival | participants will be followed for the duration of chemotherapy and for at least 1 yaer after the completation of treatment, an expected average of 18 months
  The primary efficacy endpoint is toxicity-free survival, defined as the time from randomisation up to the occurrence of related to treatment grade 2-3-4 NCI-CTCAE neurotoxicity, progression, second primary malignancy, death from any cause, whichever comes first. Subjects who have not experienced related to treatment grade 2-3-4 toxicity, and not progressed or died while on study will be censored at their last assessment date.

SECONDARY OUTCOMES:
Progression-free survival | participants will be followed for the duration of chemotherapy and for at least 1 yaer after the completation of treatment, an expected average of 18 months
  defined as the time from randomisation up to the occurrence of progression, second primary malignancy, death from any cause, whichever comes first. Subjects who have not progressed or died while on study will be censored at their last assessment date
Overall survival | participants will be followed for the duration of chemotherapy and for at least 1 yaer after the completation of treatment, an expected average of 18 months
  defined as the time from the date of randomisation to the date of death from any cause. Subjects not reported as having died at the end of the study will be censored at the date they were last known to be alive
Neuropathic pain | participants will be followed for the duration of chemotherapy and for at least 1 yaer after the completation of treatment, an expected average of 18 months
  Occurrence of neuropathic pain is defined as the presence of at least 4 of the 10 clinical signs/symptoms listed in the DN4-Questionnaire Neuropathic pain intensity is defined as the intensity of pain reported by patients (current, average and worst during the last week) during scheduled visit as assessed by a self-administered questionnaire (BPI)

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Crinò, MD, Principal Investigator — Azienda Ospedaliera di Perugia
Locations (21):
- Italy (21):
  - Istituto Oncologico del Mediterraneo, Viagrande, CT
  - Azienda Ospedaliera Ospedale S. Anna, Como
  - Azienda Ospedaliera Istituti Ospitalieri, Cremona
  - Azienda Ospedaliera di Desio e Vimercate - Presidio Ospedaliero di Desio, Desio
  - Ospedale Civile, Guastalla
  - Ospedale Alessandro Manzoni, Lecco
  - Azienda Ospedaliera Ospedale Civile di Legnano, Legnano
  - Azienda Ospedaliera Fatebenefratelli e Oftalmico, Milan
  - Istituto Europeo Di Oncologia, Milan
  - Azienda Ospedaliera San Paolo, Milan
  - Azienda Ospedaliera Ospedale San Carlo Borromeo, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione Salvatore Maugeri, Pavia
  - Azienda Ospedaliera Perugia, Perugia
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - IRCCS di Reggio Emilia, Reggio Emilia
  - Azienda Ospedaliera Busto Arsizio - Presidio Ospedaliero di Saronno, Saronno
  - Ospedale SS Annunziata - ASL1, Sassari
  - Azienda Ospedaliera Valtellina e Valchiavenna , Presidio Ospedaliero di Sondrio, Sondrio
  - Azienda Ospedaliera di Pavia, Ospedale Civile di Vigevano, Vigevano
  - Azienda Ospedaliera di Desio e Vimercate - Presidio Ospedaliero di Vimercate, Vimercate